CLINICAL TRIAL: NCT02045615
Title: Removal Wichita Fusion Nail After Knee Arthrodesis
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S56066
Record Dates: First submitted 2014-01-21; First posted 2014-01-27 (Estimated); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: Removal Wichita Fusion Nail After Knee Arthrodesis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Conventional: Conventional technique for Wichita nail extraction
- New: Proposed technique for Wichita nail extraction
  Interventions: Procedure: Proposed technique for removal of the Wichita Fusion Nail

INTERVENTIONS:
Procedure: Proposed technique for removal of the Wichita Fusion Nail
  Groups: New

SUMMARY:
The purpose of this study is to make clear how difficult it is to remove osteosynthesis materials afterwards, so surgeons will think twice before inserting intramedullary nails. Also it offers an alternative methode to remove the Wichita Fusion Nail after arthrodesis has become.

ELIGIBILITY:
Inclusion Criteria:

* Extraction of Wichita Fusion Nail

Exclusion Criteria:

* All other kinds of intramedullairy nails used to become a solid knee arhrodesis

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who had to have their Wichita Fusion Nail extracted
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Operation technique | first 4 months postop
  Was the arthrodesis site left intact? How was the Nail removed? Time for operation?

SECONDARY OUTCOMES:
Mobility | 1 year postop
Pain measurement following the Visual Analogue Scale | 1 year postop
Major complications after removal | first 2 years postop
  Amputation? Infection? Wound problems?

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Leuven, Pellenberg, Belgium